CLINICAL TRIAL: NCT06888661
Title: An Open-label, Dose-escalation Clinical Trial to Assess the Safety and Efficacy of EXG001-307 After Intrathecal Injection in Patients With Spinal Muscular Atrophy
Brief Title: Clinical Trial to Assess the Safety and Efficacy of EXG001-307 in Patients With Spinal Muscular Atrophy
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hangzhou Jiayin Biotech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EXG001-307-011
Record Dates: First submitted 2025-03-03; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Spinal Muscular Atrophy (SMA)
Keywords: SMA; AAV9; gene therapy
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation- Cohort 1 (Experimental): Dose 1 Intrathecal administration dose 1 of EXG001-307 to SMA patient (type I &type II)
  Interventions: Biological: EXG001-307 injection

INTERVENTIONS:
Biological: EXG001-307 injection — non-replicating, rAAV vector based on AAV9 containing cDNA encoding the human SMN protein.

SUMMARY:
The purpose of this trial is to evaluate safety and efficacy of intrathecal delivery of EXG001-307 as a treatment of spinal muscular atrophy .

ELIGIBILITY:
Inclusion Criteria:

1. On the day of dosing, type 1 SMA age ≤180 days, type 2 SMA age > 180 days ≤2 years, male or female.
2. Clinical history and physical signs are consistent with SMA manifestations; SMA was diagnosed by bilateral allelic SMN1 mutation (deletion or point mutation). Type 1 has 2 copies of SMN2 gene. Type 2 has ≤3 copies of SMN2 gene.

4.The subject's legal guardian understands the purpose, possible risks and interests of the study, agrees to participate in the study, completes all study procedures, tests and visits, and voluntarily signs the informed consent form.

5.During the study, the subject's legal guardian was willing to perform standard treatment requirements such as nasogastric feeding, noninvasive mechanical ventilation, and expectoration machine as recommended by the investigator.

Exclusion Criteria:

1. The presence of contraindications to lumbar puncture (including, but not limited to, signs or symptoms of skin infection at the administration site and elevated intracranial pressure), the receipt of any active intrathecal therapy, the presence of an implantable shunt tube for draining CSF, the presence of an implantable central nervous system (CSF) cannula, or any condition that interferes with CSF collection.
2. Imaging shows severe scoliosis (defined as curvature of the spine ≥ 50°).
3. Gestational age at birth was less than 35 weeks (245 days).
4. At screening, the subject had an oxygen saturation < 95% while awake or sleeping and did not receive any supplemental oxygen or respiratory support.
5. Requirement of invasive ventilation or tracheotomy, or current use of noninvasive ventilatory support for an average of ≥ 12 hours/day.
6. Weighed below the 3rd percentile by age according to the WHO Child Growth Criteria (WHO 2009).
7. Before administration, if the subject has not received or delayed vaccination according to the current month-old national vaccination plan, it will significantly affect the safety of the subject as assessed by the investigator and the medical manager of the project team;
8. Active viral infections (including HIV, hepatitis B or C seropositivity, torch virus, Epstein-Barr virus, and syphilis).
9. Serious non-respiratory disease within 2 weeks prior to screening.
10. EXG001-307 has had an upper respiratory tract infection or lower respiratory tract infection within 4 weeks prior to administration, and still has relevant clinical symptoms or is still in an unstable state of disease.
11. Other severe infections or illnesses within 4 weeks prior to administration of EXG001-307.
12. A history of bacterial meningitis or brain or spinal cord disease, including tumors, or abnormalities found on an MRI or computed tomography scan that interfere with a lumbar puncture procedure or cerebrospinal fluid circulation.
13. There are currently clinically significant heart disease or electrocardiogram abnormalities that may affect the safety assessment of subjects.
14. Known hypersensitivity to prednisolone, other glucocorticoids, or its excipients；Or cannot tolerate oral or gastrostomy tube administration of corticosteroids.
15. Immunosuppressive therapy (eg, cyclosporine, tacrolimus, methotrexate, cyclophosphamide, rituximab) other than protocol-required prophylaxis within 3 months prior to dosing.
16. Immunomodulatory drugs (eg, thymosin, interferon, etc.) are being used to treat myopathy, neuritis, diabetes mellitus (eg, immunosuppressants, glucocorticoids, insulin).
17. Prior use of other SMA therapeutic agents (e.g., nosinasenat, rispolam, and Zolgensma, etc.) or participated in clinical studies with other SMA therapeutic agents.
18. Patients with type 2 SMA who had undergone scoliosis surgery or coxopexy in the 12 months prior to screening or were scheduled to undergo scoliosis surgery or coxopexy in the next 52 weeks.
19. Major surgery is expected during study treatment.
20. Other circumstances that, in the judgment of the investigator, are not suitable for participation in this study.

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of EXG001-307 following a single intrathecal injection | up to 52 weeks after treatment
  Adverse events (AES), serious adverse events (SAEs), dose-limited toxicity types, severity, incidence, and drug relevance were evaluated after treatment.（Evaluate through examinations such as electrocardiogram, echocardiography, blood routine, blood biochemistry, coagulation function, etc. conducted during each visit）

SECONDARY OUTCOMES:
Evaluate the improvement of motor function in subjects after treatment: assessed with the BSID-III scale | up to 52 weeks after treatment
  The achievement of new milestones in the BSID-III
Evaluate the improvement of motor function in subjects after treatment: assessed with the CHOP-INTEND scale | up to 52 weeks after treatment
  Evaluate the changes in subjects' scores compared to baseline and the proportion of subjects with scores above 40 using the CHOP-INTEND scale.
Evaluate the improvement of motor function in subjects after treatment: assessed with the HINE-2 scale | up to 52 weeks after treatment
  Evaluate the achievement of motor milestones by the Hammersmith Infant Neurological Examination (HINE-2) Module 2

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghai Children's Medical Center Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The Children's Hospital of Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No